CLINICAL TRIAL: NCT00687440
Title: Pegylated Liposomal Doxorubicin (Caelyx) in Combination With Herceptin and Taxotere as First-line Chemotherapy in Metastatic Breast Cancer Patients: A 2 Stage Phase II, Open Label, Multicenter Study.
Brief Title: A Study to Determine the Activity of Caelyx With Trastuzumab and Docetaxel in the Treatment of Metastatic Breast Cancer (Study P03679)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: MDS Pharma Services (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P03679; Eudract No. 2004-003989-15
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Results first posted 2010-02-15 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Breast Neoplasm
MeSH Terms: conditions — Breast Neoplasms | interventions — liposomal doxorubicin; Docetaxel; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Caelyx, Docetaxel, Trastuzumab (Experimental): Stage 1: subjects will receive Caelyx one day every 3 weeks in combination with docetaxel one day every 3 weeks and trastuzumab once weekly during 6 cycles. At the end of this stage, based on the number of cardiac events, subjects will proceed to a second stage or restart with a lower dose of Caelyx.
  Stage 2: subjects will be treated with the recommended dose of Caelyx (defined in the first stage) in combination with docetaxel and trastuzumab.
  Interventions: Drug: Pegylated Liposomal Doxorubicin; Drug: Docetaxel; Drug: Trastuzumab

INTERVENTIONS:
Drug: Pegylated Liposomal Doxorubicin — Stage 1: 25 subjects will be treated with Caelyx IV 30 mg/m^2 on day 1, every 3 weeks
  Stage 2: 45 new patients will be treated at the recommended dose level (defined in the first step) on day 1, every 3 weeks.
  Other Names: Caelyx
Drug: Docetaxel — Stage 1 and Stage 2: Docetaxel 60 mg/m2 IV as 1-hour infusion, on day 1, every 3 weeks.
  Other Names: Taxotere
Drug: Trastuzumab — Stage 1 and Stage 2: 4 mg/kg IV 90-minute infusion loading dose. Then 2 mg/kg IV weekly during 6 cycles (18 weeks).

SUMMARY:
The purpose of this study is to evaluate, in a first stage, the safety (incidence of cardiac toxicity) of Caelyx in combination with Trastuzumab and Docetaxel; and in a second stage, the tumor response rate of this regimen. This study will be conducted in approximately 30 centers. A total of approximately 70 to 95 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

Patients must fulfill all the following criteria:

* Females aged 18 to 70 years-old.
* Willingness to participate in the study and comply with its procedures.
* Documented diagnosis of metastatic breast carcinoma (stage IV) Human Epidermal Growth Factor Receptor 2 (HER2) overexpressing (Immunohistochemistry (IHC) 3+ or Fluorescence In Situ Hybridization(FISH) +).
* No prior chemotherapy for metastatic breast cancer.
* Adjuvant or neo-adjuvant chemotherapy is allowed according to the following rules:

  * patients treated with anthracyclines if all the following conditions are met:

    * Doxorubicin total dose <= 300 mg/m^2
    * Epirubicin total dose <= 480 mg/m^2
    * Chemotherapy-free interval of > 12 months
  * no taxane-based adjuvant or neo-adjuvant chemotherapy is allowed;
  * patients treated with non-anthracycline/taxane adjuvant or neo-adjuvant chemotherapy regimens are freely eligible (i.e. cyclophosphamide/methotrexate/fluorouracil (CMF) or similar regimens).
* At least one measurable lesion according to RECIST criteria.
* Complete hematologic and biologic baseline evaluation within 2 weeks prior to start of treatment.
* Complete Tumor baseline evaluation including a total body computed tomography (CT) scan within 4 weeks prior to start of treatment.
* Left ventricular ejection fraction (LVEF) >= 50% as determined by echocardiogram or Multi Gated Acquisition (MUGA) scan.
* World Health Organization (WHO) performance status 0,1.
* Life expectancy > 3 months.
* Laboratory requirements :

  * Hematology :

    * Neutrophils > 1.5 x 10^9/L
    * Platelets > 100 x 10^9/L
    * Hemoglobin > 10 g/dL
  * Hepatic function:

    * Total bilirubin <= 1.25 x the upper-normal limits (UNL);
    * ASAT (Aspartate Aminotransferase or SGOT), ALAT (Alanine aminotransferase or SGPT) <= 2.5 x the upper-normal limits;
  * For patients with liver metastases:

    * Total bilirubin < 1.5 x the UNL (Upper limit of normal) ;
    * ASAT and/or ALAT < 3 x the UNL;
  * Renal function :

    * Serum Creatinine < 1.5 x the UNL.
* Women of child bearing potential must have a negative serum pregnancy test and be using adequate contraception.
* Patients must be accessible for treatment and follow-up.

Exclusion Criteria:

Patients will not be enrolled if any of the following criteria apply:

* Prior chemotherapy for metastatic disease.
* History of prior malignancy in the last 10 years (other than non melanoma skin cancer or excised cervical carcinoma in situ).
* Radiation to disease areas within 3 weeks of study initiation.
* Symptomatic peripheral neuropathy > grade 2 according to the National Cancer Institute (NCI) Common Toxicity Criteria.
* Other serious illness or medical condition.
* LVEF < 50% as determined by echocardiogram or MUGA scan.
* Congestive hearth failure or angina pectoris even if it is medically controlled. Previous history of myocardial infarction within 1 year from study entry, uncontrolled high risk hypertension or arrhythmia.
* History of significant neurologic or psychiatric disorders including dementia or seizures.
* Active infection.
* Active peptic ulcer, unstable diabetes mellitus or other contraindications for the use of dexamethasone.
* Concurrent treatment with other experimental drugs. Participation in another clinical trial with any investigational drug within 30 days prior to study screening.
* Concurrent treatment with corticosteroids used for reasons other than for premedication. However patients receiving chronic treatment with corticosteroids (> 6 months) at low dose (< 20 mg of methylprednisolone or equivalent dose of other corticosteroids) for whichever reason are eligible.
* Taxane-based adjuvant or neo-adjuvant chemotherapy < 12 months.
* Other concurrent chemotherapy, immunotherapy, radiotherapy or any other investigational medication, for the treatment of the tumor.
* Pregnant or breast-feeding women.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2005-07-15 (Actual); Primary Completion 2008-10-24 (Actual); Study Completion 2008-10-24 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Caelyx, Docetaxel, Trastuzumab
Started | 27 (Number of screened participants)
Completed | 15
Not Completed | 12
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 3
Not completed — Lack of Efficacy | 2
Not completed — Death | 2
Not completed — Other | 1
Not completed — Missing | 1

BASELINE CHARACTERISTICS:
Arm/Group | Caelyx, Docetaxel, Trastuzumab
Number analyzed (Participants) | 27
Age, Customized [Number; unit: years] | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 0
Region of Enrollment [Number; unit: participants]
  Italy | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had a Tumor Response, According to Standard RECIST (Response Evaluation Criteria in Solid Tumors) Criteria
Description: Those who achieved either complete (disappearance of all target lesions) or partial (at least 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD) response.
Time Frame: Week 09, Week 18, at the end of each patient's treatment, and at 3, 6, 9, and 12 months after end of treatment.
Population: Intent-to-treat population
Measure: Number; unit: Participants
Arm/Group | Caelyx, Docetaxel, Trastuzumab
Number analyzed (Participants) | 26
Participants
  Participants who had a complete tumor response | 2
  Participants who had a partial tumor response | 13
  Participants who did not have a tumor response | 11

ADVERSE EVENTS:
Arm/Group | Caelyx, Docetaxel, Trastuzumab
Serious Adverse Events (participants affected / at risk) | 6/27
Other Adverse Events (participants affected / at risk) | 21/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caelyx, Docetaxel, Trastuzumab (N=27)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
STOMATITIS (Gastrointestinal disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
MUCOSAL INFLAMMATION (General disorders) | 1 (1)
PYREXIA (General disorders) | 1 (1)
SEPSIS (Infections and infestations) | 1 (1)
EJECTION FRACTION DECREASED (Investigations) | 1 (1)
METASTASES TO MENINGES (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
COMA (Nervous system disorders) | 1 (1)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 2 (2)
HYPOTENSION (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Caelyx, Docetaxel, Trastuzumab (N=27)
LEUKOPENIA (Blood and lymphatic system disorders) | 5 (18)
LYMPHOPENIA (Blood and lymphatic system disorders) | 2 (10)
NEUTROPENIA (Blood and lymphatic system disorders) | 5 (10)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (8)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3 (6)
CONSTIPATION (Gastrointestinal disorders) | 3 (5)
DIARRHOEA (Gastrointestinal disorders) | 7 (11)
GASTRITIS (Gastrointestinal disorders) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 8 (9)
STOMATITIS (Gastrointestinal disorders) | 7 (28)
VOMITING (Gastrointestinal disorders) | 3 (3)
ASTHENIA (General disorders) | 8 (10)
CHEST PAIN (General disorders) | 2 (5)
FATIGUE (General disorders) | 2 (3)
MUCOSAL INFLAMMATION (General disorders) | 6 (22)
OEDEMA PERIPHERAL (General disorders) | 2 (3)
PYREXIA (General disorders) | 6 (7)
HEADACHE (Nervous system disorders) | 2 (2)
PARAESTHESIA (Nervous system disorders) | 3 (3)
ALOPECIA (Skin and subcutaneous tissue disorders) | 4 (4)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 2 (2)
ONYCHOLYSIS (Skin and subcutaneous tissue disorders) | 2 (2)
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 16 (43)
RASH (Skin and subcutaneous tissue disorders) | 3 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No